CLINICAL TRIAL: NCT00447577
Title: A Clinical Safety and Efficacy Evaluation of Zylet (Loteprednol Etabonate and Tobramycin Ophthalmic Suspension) vs. Tobradex (Tobramycin and Dexamethasone Ophthalmic Suspension) in the Treatment of Blepharokeratoconjunctivitis
Brief Title: Zylet vs TobraDex in Blepharokeratoconjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 512
Record Dates: First submitted 2007-03-12; First posted 2007-03-14 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Blepharokeratoconjunctivitis
MeSH Terms: interventions — Loteprednol Etabonate; Tobramycin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zylet (Experimental): Loteprednol etabonate and tobramycin ophthalmic suspension, 0.5%/0.3% (Zylet)
  Interventions: Drug: Loteprednol etabonate and tobramycin ophthalmic suspension
- Tobradex (Active Comparator): Tobradex (tobramycin and dexamethasone ophthalmic suspension, 0.3%/0.1%), US marketed product (Alcon) from commercial lots.
  Interventions: Drug: Tobramycin and dexamethasone ophthalmic suspension

INTERVENTIONS:
Drug: Loteprednol etabonate and tobramycin ophthalmic suspension — Subjects will self-administer the study drug in the affected eye(s) 4 times a day (QID) for 14 days.
  Arms: Zylet
Drug: Tobramycin and dexamethasone ophthalmic suspension — Subjects will self-administer the study drug in the affected eye(s) 4 times a day (QID) for 14 days.
  Arms: Tobradex

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of Zylet vs. Tobradex in the treatment of ocular inflammation associated with blepharokeratoconjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Must be able and willing to comply with all treatment and follow up procedures
* Must have the ability to understand and sign an Informed Consent Form and provide Health Insurance Portability and Accountability Act (HIPAA) authorization
* Must be able to self-administer drugs
* Must have a clinical diagnosis of blepharokeratoconjunctivitis in at least one eye (total Ocular Signs and Symptoms score of at least 10, with at least one ocular sign and one ocular symptom each having a score of Grade 2 level or higher)
* Women of childbearing potential must be sexually inactive or using an approved birth control methods and must have a negative urine pregnancy test
* Must be willing to discontinue contact lens use for the duration of the study
* Must have pin-holed Snellen visual acuity equal to or better than 20/40 in both eyes

Exclusion Criteria:

* Any uncontrolled systemic disease or debilitating disease (e.g. cardiovascular disease, hypertension, diabetes, or cystic fibrosis)
* Known hypersensitivity to the study drugs or their components (including benzalkonium chloride) or contraindications to tobramycin or ocular corticosteroids
* Use of any systemic or topical ophthalmic non-steroidal anti-inflammatory agents, analgesics, and antihistamines that cannot be discontinued during the study
* Use of any topical ophthalmic medications, including tear substitutes, within 2 hours before and that cannot be discontinued during the study
* Use of any systemic or topical ophthalmic antibiotic agents within 72 hours before and that cannot be discontinued during the study
* Use of any systemic or topical ophthalmic corticosteroid agents within 7 days before and that cannot be discontinued during the study
* Use of any systemic or topical ophthalmic mast cell stabilizers within 14 days before and that cannot be discontinued during the study
* Use of any topical ophthalmic immunosuppressant (e.g. Restasis) agents within 30 days before and that cannot be discontinued during the study
* Suspected preseptal cellulites, or any other disease conditions which the Investigator determines could interfere with the safety and efficacy evaluations of the study drug
* Suspected dacrocystitis
* Participation in an ophthalmic drug or device research study within the 30 days prior to entry in this study
* Ocular surgery (including laser surgery) in either eye within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2007-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint for this study is the change from baseline to Day 15 in the signs and symptoms composite score | 15 days

SECONDARY OUTCOMES:
The distribution of Investigator global assessment at each visit. | Visit 2, 3 & 4
The percentage of eyes that were considered improved or cured at each visit based on the Investigator global assessment. | Visit 2, 3 & 4
The change from baseline to Day 7 (Visit 3) and to Day 3 (Visit 2) in the signs and symptoms composite score. | Visit 2 & 3
The change from baseline to each visit in the signs composite score and the symptoms composite score. | Visit 1, 2, 3 & 4
The change from baseline to each visit in the Blepharitis signs composite score, the conjunctivitis signs composite score, and the Keratitis signs composite score. | Visit 1, 2, 3 & 4
The change from baseline to each visit in individual signs and symptoms. | Visit 1, 2, 3 & 4
VA, Biomicroscopy, and IOP assessments at each visit | Visit 1, 2, 3 & 4
Adverse Events | Visit 1, 2, 3 & 4

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Comstock, OD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Cornerstone Eye Care, High Point, North Carolina, United States

REFERENCES:
- [Derived] White EM, Macy JI, Bateman KM, Comstock TL. Comparison of the safety and efficacy of loteprednol 0.5%/tobramycin 0.3% with dexamethasone 0.1%/tobramycin 0.3% in the treatment of blepharokeratoconjunctivitis. Curr Med Res Opin. 2008 Jan;24(1):287-96. doi: 10.1185/030079908x253898. PMID 18062846